CLINICAL TRIAL: NCT06283602
Title: Erosive Tooth Wear, Caries Experience and Periodontal Health in Children and Adolescents With Obesity and Normal Weight
Brief Title: Oral Health in Children and Adolescents With Obesity and Normal Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aslı Sogukpınar, Assistant Professor, Mersin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/17
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pediatric Obesity; Pediatric Dentistry
Keywords: dental caries; periodontal health; children; obesity; erosive tooth wear
MeSH Terms: conditions — Pediatric Obesity; Dental Caries; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kahramanmaraş Sütçü İmam University (Other): Patient who apply to our clinic for routine paediatric treatment for the included in the study
  Interventions: Diagnostic Test: oral health status

INTERVENTIONS:
Diagnostic Test: oral health status — the dentists examined the dried teeth with a probe and mount mirror in a dental unit.

SUMMARY:
We aimed to compare the oral health status (dmft/DMFT index, IDCAS-II, BEWE, plaque index, gingival index, probing depth) between normal-weight (NW) and obese (OW) children/adolescents.

82 participants aged 6-16 years were concluded in this cross-sectional study. The children/adolescents were classified according to the body mass index (BMI): NW (n=41) and OW (n=41). Caries experience was assessed by the International Caries Detection and Assessment System (ICDAS-II), decay, missing, filling teeth (dmft) for the primary teeth and (DMFT) for the permanent teeth, erosive tooth wear using Basic Erosive Wear Examination (BEWE), Plaque Index (PI) and Gingival Index (GI), Probing Depth (PD).

DETAILED DESCRIPTION:
Also, the relationship between procalcitonin (PCT), C-reactive protein (CRP), parathormone (PTH), and 25(OH)D blood biochemistry and oral health was evaluated in obese children/adolescents.

ELIGIBILITY:
Inclusion Criteria: 6-16 years obesity children and adolescents

* 6-16 years healthy children and adolescents

Exclusion Criteria:

* Infection,
* diabetes, leukemia, asthma, bronchitis, cognitive neuromotor disorder, hormonal disease

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
the results of DMFT, plaque and gingival indies | 12 months
  The results of the study indicate that individuals with obesity tend to exhibit significantly higher scores for DMFT, plaque, and gingival index as compared to those with normal weight t significantly higher scores for DMFT, plaque, and gingival index as compared to those with normal weight (p<0.05)
the results of dmft, BEWE, ICDAS-II, probing dept | up to 12 months
  No significant difference was observed concerning dmft and other factors (p>0.05)
Comparison of demographic attributes between obese and normal weights | 12 months
  Significant disparities were identified between patients with normal weight and those who were obese, particularly in BMI, income, and tooth brushing habits. Obese patients exhibited considerably higher BMI scores in comparison to those with normal weight (p<0.001).Body mass index (BMIs; kg/m2) was calculated by the pediatrician using the patients' height (meters) and weight (kilograms). BMI 5-85th percentile normal weight according to gender and age; BMI 85- 95 percentile overweight; Those at the 95th percentile and above were considered obese

SECONDARY OUTCOMES:
biochemical parameters of obese individuals | 11 months
  Procalcitonin exhibited significantly negative correlation between DMFT and ICDAS-II (p<0.05).
other biochemical parameters of obese individuals | up to 11 months
  No significant correlation was found between the biomarkers and other investigated factors (p>0.05)

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Soğukpınar Önsüren, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided